CLINICAL TRIAL: NCT06214403
Title: Antimicrobial Resistant Organism Decolonization After Microbiome Perturbation (ARO-DECAMP): a Multi-centre, Randomized, Placebo-controlled Feasibility Pilot Trial
Brief Title: Antimicrobial Resistant Organism Decolonization After Microbiome Perturbation
Acronym: ARO-DECAMP
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-5419
Record Dates: First submitted 2023-12-21; First posted 2024-01-19 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Gram-negative Bacteremia; Microbial Colonization; Antibiotic Resistant Infection
Keywords: Microbial consortia; Microbiome; Decolonization; Infection; Bacteremia; Antibiotic; Microbiota; Antibiotic resistance
MeSH Terms: conditions — Communicable Diseases; Infections; Bacteremia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MET-2 (Experimental): Participants randomized to the intervention will receive MET-2 daily for 10 days. MET-2 capsules are administered orally at 0.5 g per capsule, containing 3.1 x 10^5-10^11 colony forming units (CFU). An initial loading dose of 10 MET-2 capsules/day will be taken for 2 days (5 grams total). For the following 8 days, participants will take a maintenance dose of 3 MET-2 capsules/day (1.5 grams total).
  Interventions: Drug: MET-2
- Placebo (Placebo Comparator): Participants randomized to the placebo will receive microcrystalline cellulose in a capsule, identical in appearance to MET-2 but not containing live bacteria. Participants will take the placebo in the same dosing schedule as the MET-2 arm: 10 capsules daily for 2 days, followed by 3 capsules daily for 8 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MET-2 — Microbial Ecosystem Therapeutics (MET) is a defined microbial community derived from healthy donor stool. MET capsules are orally administered mixtures of pure cultures of human-derived bacterial strains.
  Arms: MET-2
Drug: Placebo — Microcrystalline Cellulose
  Arms: Placebo

SUMMARY:
ARO-DECAMP is a multi-centre, placebo-controlled, pilot and feasibility randomized controlled trial for the microbial consortium Microbial Ecosystem Therapeutic-2. Non-intensive care unit patients ≥ 18 years old diagnosed with a bloodstream infection and receiving treatment for an antibiotic resistant organism will be included. Participants will be randomized to receive either MET-2 or placebo for 10 days. Recruitment rate and study intervention adherence will be evaluated for feasibility. Participants will be followed for 180 days, and biological samples will be collected periodically for clinical, ecological, and biomarker outcomes.

DETAILED DESCRIPTION:
Reconstituting the perturbed microbiome is a novel therapeutic modality with the potential to decrease ARO colonization and infection and combat AMR without additional pressure for selection of further antimicrobial resistance. No trial has yet assessed the potential of a therapeutic microbial consortium for ARO decolonization and infection prevention after antibiotic treatment.

The investigational product, Microbial Ecosystem Therapeutic-2 (MET-2), is a defined microbial community derived from healthy donor stool. MET capsules are orally administered mixtures of bacterial strains cultured from the stool of a healthy donor. This study is designed to determine if a trial of administration of MET-2 after antibiotic treatment for bloodstream infections is feasible. Stool and plasma biomarkers to assess the effects of the intervention will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) inpatient not admitted to the ICU or equivalent (step-up and step-down units are eligible)
2. Positive blood culture with an ARO:

   * AmpC beta-lactamase producing species: Enterobacter cloacae, Citrobacter spp., Klebsiella aerogenes, Serratia spp., Morganella morganii, Hafnia alvei OR
   * ESBL-producing gram-negative bacilli
3. Currently receiving treatment for the bloodstream infection

Exclusion Criteria:

1. Inability to swallow oral MET-2 or placebo capsule
2. Recipient of small bowel transplant
3. Inflammatory bowel disease, short bowel syndrome, diverting/non-diverting ileo/colostomy
4. Use of >3 days over-the-counter or prescription probiotics (not including food additives) within 10 days of enrolment
5. Receipt of fecal microbiota transplant (FMT) within 3 months of enrolment
6. Absolute neutrophil count <0.5x109/L
7. Death expected within 72 hours of enrolment
8. Planned continuation of non-prophylaxis antimicrobial therapy active against the bloodstream isolate for >42 days
9. Known pregnancy, planning to become pregnant during the study period, or breastfeeding
10. Any other reason in view of the site investigator or treating team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate overall and by study site | 1.5 years
  Defined by the numbers of eligible, consented, and randomized patients
Adherence to MET-2/placebo for the treatment duration | 30 days
  Defined as >80% of loading dose (16/20 pills) + >75% of daily doses (18/24 pills) for the maintenance period, as determined by returned unused capsules

SECONDARY OUTCOMES:
Change in microbiome composition after intervention | 180 days
  Assessment of gut microbiome composition in pre- and post-randomization stool samples using bacterial culture and culture-independent (sequencing) assays.
Number of biomarker samples collected, by sample type and timepoint | 30 days
  Successful adherence to biomarker sample collection is defined as >80% of participants having samples suitable for analysis at 30 days post-intervention
Concentration of potential biomarkers in pre- and post-randomization blood and urine samples | 180 days
  Microbial-derived metabolites (short chain fatty acids and bile acids in blood, and 3-indoxyl sulfate in urine), markers of intestinal permeability (soluble CD14, LPS, LPS-binding protein, ZO-1, intestinal fatty acid protein), immune cell profiles (CD8 T lymphocytes, CD4 T lymphocytes, T regulatory cells, B lymphocytes, Th17 cells, Th1 cells).

OTHER OUTCOMES:
Adverse events | 180 days
  Frequency and grade
90- and 180-day infection rate | 180 days
  Infection will be defined as either isolation of a pathogenic species from any sterile site OR the initiation of a therapeutic course of antimicrobials with or without isolation of a pathogenic species from a sterile or non-sterile site
ARO colonization by culture at 30 and 90 days post-intervention | 90 days
  Defined as any positive result for ARO from any site
Determine 90- and 180-day recurrence/re-infection rates (with the same organism) in each treatment arm | 180 days
AMR gene complement by sequencing at 30 and 90 days post-intervention | 90 days
90- and 180-day all-cause mortality | 180 days
ICU and hospital lengths of stay | 180 days
C. difficile carriage at days 30 and 90 | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Coburn, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (4):
- Canada (4):
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Sinai Health, Toronto, Ontario